CLINICAL TRIAL: NCT01894165
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled, Single-Dose, Sequential-Cohort, Dose-Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ALXN1101 in Healthy Adult Subjects
Brief Title: Phase 1 Single Dose Study of ALXN1101 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Origin Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALXN1101-MCD-101
Record Dates: First submitted 2013-06-27; First posted 2013-07-10 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Molybdenum Cofactor Deficiency (MoCD); Rare Autosomal Recessive Disorder; Deficiency of Activity of Molybdenum-dependent Enzymes (Sulfite Oxidase [SOX], Xanthine Dehydrogenase, and Aldehyde Oxidase)
Keywords: molybdenum cofactor deficiency (MoCD); deficiency of activity of molybdenum-dependent enzymes
MeSH Terms: conditions — Molybdenum cofactor deficiency | interventions — nulibry

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALXN1101 (Experimental): Four cohorts planned. Within each cohort, healthy volunteers are randomized to ALXN1101 IV single dose or placebo IV single dose. Each subsequent cohort is testing an increased dose of ALXN1101 IV or placebo IV.
  Interventions: Drug: ALXN1101
- Placebo (Placebo Comparator): Four cohorts planned. Within each cohort, healthy volunteers are randomized to ALXN1101 IV single dose or placebo IV single dose. Each subsequent cohort is testing an increased dose of ALXN1101 IV or placebo IV.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALXN1101 — Randomized to receive a single dose of ALXN1101 or placebo as per assigned cohort dose level.
  Arms: ALXN1101
Drug: Placebo — Randomized to receive a single dose of ALXN1101 or placebo as per assigned cohort dose level.
  Arms: Placebo

SUMMARY:
Phase 1 single dose study of ALXN1101 in healthy volunteers.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), randomized, blinded, placebo-controlled, single-dose, sequential-cohort, dose-escalation study to evaluate the safety, tolerability, and pharmacokinetics (PK) of a single dose of ALXN1101 in healthy adult subjects.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female subjects ≥ 18 and ≤ 60 years of age and weight ≥ 55 kg and ≤ 100 kg
2. Willing and able to give written informed consent
3. Female subjects of child bearing potential must have a negative serum pregnancy test or must be practicing an approved contraceptive regimen for the duration of the study
4. Male subjects must be practicing an acceptable barrier method of contraception

Key Exclusion Criteria:

1. Pregnant or nursing female subjects
2. QTcF > 450 msec for males and > 470 msec for females, or a family history of Long QT Syndrome.
3. CrCl < 80 mL/min
4. CBC in acceptable range; SGOT or SGPT above the ULN
5. HIV, Hepatitis B or Hepatitis C virus infection
6. Other active systemic infection or malignancy
7. Investigational drug study within 60 days
8. Major surgery within the prior 90 days
9. History of illicit drug use or chronic alcohol dependence within 2 years prior to this study
10. Positive urine drug toxicology screen or serum alcohol test
11. Alcohol consumption within 48 hours prior to study drug administration
12. Recently donated or lost ≥ 499 mL of blood
13. Recent hormone replacement therapy or use of prescription medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single dose of ALXN1101 in healthy adult subjects | following the Day 30 visit for the last study subject
  Physical examination, vital signs, ECGs, laboratory evaluations, and Adverse Events.

SECONDARY OUTCOMES:
PK parameters of ALXN1101 | following the Day 5 visit for the last study subject
  PK parameters of ALXN1101 will be estimated including, but not limited to,maximum observed plasma concentration (Cmax), time to maximum observed plasma concentration (tmax), terminal elimination halflife (t½), area under the plasma concentration-time curve (AUC), total body clearance (CL), and volume of distribution (Vd).

OTHER OUTCOMES:
Exploratory biochemical marker assessments | following the Day 30 visit for the last study subject
  To evaluate urine, serum or plasma concentrations of biochemical markers including S-sulfocysteine, xanthine, uric acid, creatinine, and other exploratory biochemical markers.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MD, Principal Investigator — Parexel Baltimore Early Phase Clinical Unit
Locations (1):
- Parexel Baltimore EPCU, Baltimore, Maryland, United States